CLINICAL TRIAL: NCT00165295
Title: Phase II Study of Sildenafil Citrate in Waldenstrom's Macroglobulinemia
Brief Title: Sildenafil Citrate in Waldenstrom's Macroglobulinemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: Beth Israel Deaconess Medical Center (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 05-087
Record Dates: First submitted 2005-09-09; First posted 2005-09-14 (Estimated); Last update posted 2011-06-27 (Estimated); Status verified 2011-06

CONDITIONS: Waldenstrom's Macroglobulinemia
Keywords: sildenafil citrate; Viagra; Waldenstrom's macroglobulinemia
MeSH Terms: conditions — Waldenstrom Macroglobulinemia | interventions — Sildenafil Citrate

INTERVENTIONS:
Drug: Sildenafil citrate (Viagra)

SUMMARY:
The purpose of this study is to determine the effects (good or bad) that sildenafil (Viagra) has on patients with slow growing Waldenstrom's macroglobulinemia (WM). Sildenafil blocks the function of several proteins necessary to the survival of certain types of cancer and laboratory tests have shown that it can destroy WM cells.

DETAILED DESCRIPTION:
* Sildenafil will be given orally (at home) at a reduced dose for the first week, then each week for 3 more weeks, the dose will be increased. If the patient has no major side effects, then they will receive the maximal dose for 2 years. If they have major side effects, then the dose of the drug might be lowered or the drug stopped.
* Sildenafil will be continued until their is disease progression or serious side effects.
* While patients are receiving sildenafil, they will be seen in the clinic on months 1,2,9,15 and 21 for blood tests and a subject questionnaire. They will also be seen on months 3,6,12,18 and 24 for a physical exam, blood test, physical assessment test, CT scans of chest, abdomen and pelvis, and a subject questionnaire.
* At the end of the study (month 24) a physical exam, blood tests, physical assessment test and a questionnaire will be conducted.
* Follow-up includes clinic visits at month 27,33,39 and 45 for blood tests and a questionnaire as well as visits at month 30,36,42 and 48 for physical exam, blood tests, physical assessment test, bone marrow aspirate and biopsy, CT scans of chest, abdomen and pelvis, and a questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* Clinicopathological diagnosis of Waldenstrom's macroglobulinemia
* Measurable disease, defined as presence of immunoglobulin M (IgM) paraprotein with a minimum IgM level of > 2 times the upper limit of each institution's normal value
* Slowly progressing disease not requiring therapy for at least 3-6 months
* ECOG performance status 0,1 or 2
* Total bilirubin < 2 x ULN
* SGOT < 3 x ULN
* Creatinine < 2 x ULN

Exclusion Criteria:

* Pregnant or breast-feeding women
* Patients who are using organic nitrates or alpha-blockers
* Grade III/IV cardiac problems
* Resting hypotension (BP < 90/50) or hypertension (BP > 170/110)
* Cardiac failure or coronary artery disease causing unstable angina
* Evidence of left ventricular outflow obstruction
* Impaired autonomic control of blood pressure
* Sickle cell anemia
* History of priapism
* Severe and/or uncontrolled medical disease
* Known chronic liver disease
* Currently using ritonavir
* History of retinal pigmentosa

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30
Dates: Start 2005-09; Primary Completion 2007-06 (Actual); Study Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
To determine response, time to progression and safety for sildenafil citrate therapy in patients with slowly progressing Waldenstrom's macroglobulinemia.

CONTACTS AND LOCATIONS:
Overall Officials: Steven P. Treon, MD, MA, PhD, Principal Investigator — Dana-Farber Cancer Institute
Locations (1):
- Dana-Farber Cancer Institute, Boston, Massachusetts, United States